CLINICAL TRIAL: NCT07236164
Title: Effectiveness of the Guided Self-Help CBT Manual 'Khushi or Khatoon (KoK)' in Cancer Patients: A Randomised Controlled Trial
Brief Title: Effectiveness of a Guided Self-Help CBT Manual 'KOK' in Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Association of Cognitive Therapists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RCTCANCER2025
Record Dates: First submitted 2025-09-25; First posted 2025-11-19 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Depression; Anxiety; Cancer
Keywords: Depression; Anxiety; Guided self-help; Cancer; CBT
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial with two parallel groups: an intervention group receiving the CBT self-help manual and a control group receiving usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally adapted guided self-help CBT manual 'Khushi or Khatoon (KoK)' (Experimental): Participants will receive the culturally adapted Guided self-help CBT manual 'Khushi or Khatoon (KoK)'. The manual includes eight modules on managing anxiety and depression. The modules focus on cognitive restructuring, problem solving, behavioural activation, conflict management, interpersonal relationships, mental health and well-being, and self-care. Each module is delivered over one week. The intervention uses culturally appropriate stories, drawings, and examples from local folklore and religious contexts to describe the concepts of CBT.
  Interventions: Behavioral: Culturally adapted guided self-help CBT manual 'Khushi or Khatoon (KoK)'
- Treatment as Usual (No Intervention): Receive usual care, which may include standard support provided by the oncology team.

INTERVENTIONS:
Behavioral: Culturally adapted guided self-help CBT manual 'Khushi or Khatoon (KoK)' — Participants will receive the culturally adapted guided self-help CBT manual 'Khushi or Khatoon (KoK)'. The manual includes eight modules on managing anxiety and depression. The modules focus on cognitive restructuring, problem solving, behavioural activation, conflict management, interpersonal relationships, mental health and well-being, and self-care. Each module is delivered over one week. The intervention uses culturally appropriate stories, drawings, and examples from local folklore and religious contexts to describe the concepts of CBT.
  Arms: Culturally adapted guided self-help CBT manual 'Khushi or Khatoon (KoK)'

SUMMARY:
This study aimed to assess the feasibility, acceptability, and preliminary efficacy of the Guided self-help CBT intervention 'Khushi or Khatoon' to treat anxiety and depression, and enhance quality of life and satisfaction with treatment in cancer patients.

DETAILED DESCRIPTION:
Cancer diagnosis and treatment are profoundly distressing experiences that can lead to significant psychological challenges, including depression, anxiety, and fear of recurrence. These psychological issues not only affect the quality of life of cancer patients but can also interfere with their physical health, treatment adherence, and overall recovery.

Cognitive Behavioural Therapy (CBT) is an evidence-based psychological intervention that has been widely recognised for its effectiveness in managing anxiety and depression in various patient populations, including cancer patients. CBT focuses on identifying and changing negative thought patterns and behaviours that contribute to emotional distress. However, access to skilled therapists may be limited, especially in resource-constrained settings, or for patients who are unable to attend in-person sessions due to their condition or logistical issues.

Various CBT-based self-help programs are effective in the West (Cuijpers, 1997; Gould and Clum, 1993; Marrs, 1995; Scogin et al., 1990). However, CBT requires a person to be literate, especially for guided self-help or self-help. Pakistan has a literacy rate (ability to read or write) of 58%. An estimated 67% of children study up to primary level (years 1-5), and an estimated 43% have achieved secondary education (up to year 12). These are mostly people from low socio-economic backgrounds who are less likely to suffer from mental health problems such as depression and anxiety.

A Guided self-help CBT manual, based on the core principles of CBT, could provide an accessible, cost-effective way to support cancer patients in managing their psychological distress. This study aims to evaluate the effectiveness of such a self-help manual in reducing symptoms of anxiety, depression, and overall psychological distress among cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years)
* Clinical diagnosis of cancer
* Experiencing moderate to severe psychological distress (HADS score ≥ 8)
* Able to read and write the Urdu language
* Willing to participate and provide informed consent

Exclusion Criteria:

* Severe psychiatric conditions requiring immediate intervention/hospitalisation
* Cognitive impairments preventing understanding of the manual/therapy
* Visual impairments that may prevent the reading of the manual
* Already been receiving any psychological therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Preliminary efficacy of Guided self-help CBT manual 'Khushi or Khatoon' in treating depression and anxiety in cancer patients | 8 weeks
  By comparing pre- and post-therapy depression and anxiety scores using the Hospital Anxiety and Depression Scale. The scale has a score range of 0-21 with a cut off of 8, higher scores indicate clinically significant depression/anxiety. A low post-treatment score on the Hospital Anxiety and Depression Scale is the desired outcome.
Feasibility of the Guided Self-Help CBT manual 'Khushi or Khatoon' for depressed and anxious cancer patients | 8 weeks
  By using indicators like recruitment success, dropout rates, and completion rates recorded in numbers during study
Acceptability of the Guided Self-Help CBT manual 'Khushi or Khatoon' in depressed and anxious cancer patients | 8 weeks
  Assessed through patients' satisfaction using the Verona satisfaction scale. An average score on the scale ranges from 1-5. High score on the scale indicates more satisfaction with the treatment and thus is the desired outcome.

SECONDARY OUTCOMES:
Quality of life of cancer patients | 8 weeks
  By comparing pre- and post-therapy scores on the World Health Organization Disability Assessment Schedule. The average score on the scale ranges from 0-4. Low score indicates less decline in functioning. Thus, decreased post-assessment scale score is the desired outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Farooq Naeem, Principal Investigator — Professional Association of Cognitive Therapy
Locations (1):
- Pakistan Association of Cognitive Therapists, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No